CLINICAL TRIAL: NCT04895176
Title: incidenCe and predictOrs of heaRt fAiLure After Acute coronarY Syndrome: CORALYS
Acronym: CORALYS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, Principal Investigator, A.O.U. Città della Salute e della Scienza
Other Study IDs: CORALYS
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Acute Coronary Syndrome; Heart Failure
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single-cohort retrospective study evaluating the incidence and prognostic markers of heart failure following acute coronary syndrome treated by percutaneous coronary intervention

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is the most common cause of heart failure (HF) world-wide. Primary percutaneous coronary intervention (PCI) has deeply improved short and long-term survival after ACS, but his impact on incidence of downstream heart failure still remains unclear and heart failure after ACS represents the major driver of late morbidity, mortality and healthcare cost.

Many predictors and determinant of heart failure after MI have been evaluated, however, to date, the optimal combination of parameters to predict heart failure after MI needs to be defined and very little is known about the prognostic markers in unstable angina setting

The aim of this retrospective study:

* to show the incidence of heart failure after acute coronary artery syndrome, and the relation between the type of ACS and following incidence of HF.
* to clarify which features could be routinely identified as prognostic markers. This study is a multi-center non-randomized, single-cohort retrospective study including consecutive patients with acute coronary syndrome treated by percutaneous coronary intervention between 2017 and 2019, without known previous heart failure (baseline EF > 40% and no medical therapy with loop diuretics), with at least 12 months of follow-up.

It is possible to anticipate that the main findings of the present study will fill fundamental knowledge gaps regarding incidence of heart failure following coronary events.

Among this, the study could suggest specific clinical and epidemiological features related to the risk of development of HF, leading to a better medical treatment and reducing risk for further hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* • Informed consent

  * Age ≥ 18 years
  * Previous acute coronary syndrome with percutaneous coronary revascularization
  * Baseline EF > 40%
  * At least 12 months of follow-up

Exclusion Criteria:

* • Significant valvular heart disease (greater than mild stenosis or moderate regurgitation) before ACS

  * Type 1, 3, 4, 5 pulmonary hypertension (14) before ACS
  * Constrictive pericarditis before ACS
  * Primary or infiltrative cardiomyopathies
  * Heart transplantation
  * Medical therapy with loop diuretics for heart failure before ACS
  * Previous hospitalizations for heart failure or clinical sign of heart failure detected outpatient before ACS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with acute coronary syndrome treated by percutaneous coronary intervention between 2017 and 2019, without known previous heart failure (baseline EF > 40% and no medical therapy with loop diuretics), with at least 12 months of follow-up
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Heart Failure after Acute Coronary Artery Syndrome | 12 month
  To show the incidence of heart failure after acute coronary artery syndrome.
Identify prognostic markers | 12 month
  To clarify which features could be routinely identified as prognostic markers in this setting

SECONDARY OUTCOMES:
The relation between the type of ACS and incidence of HF | 12 month
  the relation between the type of ACS and following incidence of HF will be investigated

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio D'Ascenzo, MD, Principal Investigator — AOU Città della salute e della Scienza
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy

REFERENCES:
- [Derived] D'Ascenzo F, Fabris E, DeGregorio C, Mittone G, De Filippo O, Wanha W, Leonardi S, Roubin SR, Chinaglia A, Truffa A, Huczek Z, Gaibazzi N, Ielasi A, Cortese B, Borin A, Pagliaro B, Nunez-Gil IJ, Ugo F, Marengo G, Barbieri L, Marchini F, Desperak P, Melendo-Viu M, Montalto C, Bianco M, Bruno F, Mancone M, Ferrandez-Escarabajal M, Morici N, Scaglione M, Tuttolomondo D, Gasior M, Mazurek M, Gallone G, Campo G, Wojakowski W, Abu Assi E, Stefanini G, Sinagra G, de Ferrari GM. Forecasting the Risk of Heart Failure Hospitalization After Acute Coronary Syndromes: the CORALYS HF Score. Am J Cardiol. 2023 Nov 1;206:320-329. doi: 10.1016/j.amjcard.2023.08.010. Epub 2023 Sep 19. PMID 37734293
- [Derived] Bruno F, Marengo G, De Filippo O, Wanha W, Leonardi S, Raposeiras Roubin S, Fabris E, Popovic M, Giannino G, Truffa A, Huczek Z, Gaibazzi N, Ielasi A, Cortese B, Borin A, Nunez-Gil IJ, Melis D, Ugo F, Bianco M, Barbieri L, Marchini F, Desperak P, Montalto C, Melendo-Viu M, Elia E, Mancone M, Buono A, Ferrandez-Escarabajal M, Morici N, Scaglione M, Tuttolomondo D, Sardella G, Gasior M, Mazurek M, Gallone G, Campo G, Wojakowski W, Abu-Assi E, Sinagra G, De Ferrari GM, D'Ascenzo F; Collaborators. Impact of Complete Revascularization on Development of Heart Failure in Patients With Acute Coronary Syndrome and Multivessel Disease: A Subanalysis of the CORALYS Registry. J Am Heart Assoc. 2023 Aug;12(15):e028475. doi: 10.1161/JAHA.122.028475. Epub 2023 Jul 25. PMID 37489724